CLINICAL TRIAL: NCT01456897
Title: A Long-term Trial of OPC-34712 in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 331-10-003; JapicCTI-111632 (Other: JAPIC)
Record Dates: First submitted 2011-10-11; First posted 2011-10-21 (Estimated); Results first posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2016-10

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OPC-34712 (Experimental)
  Interventions: Drug: OPC-34712

INTERVENTIONS:
Drug: OPC-34712 — orally administered once daily

SUMMARY:
To investigate the safety and efficacy of long-term administration of OPC-34712 in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 years or older (at time of informed consent) diagnosed with schizophrenia based on DSM-IV-TR diagnostic criteria
* Outpatients who are receiving an oral antipsychotic treatment (other than clozapine), who are considered to require maintenance therapy using antipsychotics, and for whom monotherapy with OPC-34712 is considered feasible

Exclusion Criteria:

* Female patients who are breastfeeding or who have a positive pregnancy test (urine) result prior to receiving investigational medicinal product
* Patients who are diagnosed with a disease other than schizophrenia (schizoaffective disorder, major depressive disorder, bipolar disorder, posttraumatic stress disorder, anxiety disorder, delirium, dementia, amnesia, or other cognitive disorder) based on current DSM-IV-TR Axis Ι criteria, or who are diagnosed with a personality disorder (borderline, paranoid, histrionic, schizotypal, schizoid, or antisocial)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2011-10; Primary Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyoji Imaoka, Operating Officer, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Kanto Region, Japan

REFERENCES:
- [Derived] Ishigooka J, Usami T, Iwashita S, Kojima Y, Matsuo S. Post-hoc analysis investigating the safety and efficacy of brexpiprazole in Japanese patients with schizophrenia who were switched from other antipsychotics in a long-term study (Secondary Publication). Neuropsychopharmacol Rep. 2020 Jun;40(2):122-129. doi: 10.1002/npr2.12107. Epub 2020 Apr 15. PMID 32297486

RESULTS

PARTICIPANT FLOW:
Groups:
- New Subjects: Participants who had not previously participated in a brexpiprazole clinical study and who received 1-4 mg of daily treatment with open label brexpiprazole in this trial
- Rollover Subjects: Participants who rolled over from, and received blinded brexpiprazole or placebo in the randomized, double-blind, placebo-controlled Phase 2/3 efficacy studies (331-10-002); all received 1-4 mg of daily treatment with open label brexpiprazole in this trial
Period: Overall Study
Arm/Group | New Subjects | Rollover Subjects
Started | 184 | 98
Completed | 109 | 41
Not Completed | 75 | 57
Not completed — Adverse Event | 19 | 22
Not completed — Protocol Violation | 3 | 4
Not completed — Physician Decision | 5 | 3
Not completed — Withdrawal by Subject | 44 | 17
Not completed — Lack of Efficacy | 4 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | New Subjects | Rollover Subjects | Total
Number analyzed (Participants) | 184 | 98 | 282
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 155 | 98 | 253
  >=65 years | 29 | 0 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (14.7) | 42.5 (12.5) | 44.4 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 58 | 152
  Male | 90 | 40 | 130
Region of Enrollment [Number; unit: participants]
  Japan | 184 | 98 | 282

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events
Description: A treatment-emergent adverse event (TEAE) is defined as an AE that started after start of investigational medicinal product (IMP) treatment.
Time Frame: From Baseline up to 52 Weeks
Population: Safety sample included those participants who had treated IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | New Subjects | Rollover Subjects
Number analyzed (Participants) | 183 | 98
Participants
  Treatment-Emergent Adverse Events (TEAE) | 156 | 79
  Potentially Drug-related TEAE | 95 | 38
  Death | 0 | 0
  SAE | 19 | 18
  Severe Treatment-Emergent Adverse Event | 8 | 7
  Discontinued Due to Adverse Events | 20 | 23

2. Secondary Outcome: Mean Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: The PANSS consisted of 3 subscales with 30 symptom constructs (positive subscale (7): delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/perseckion, and hostility; negative subscale (7): blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity and conversation flow, stereotyped thinking and general psychopathology subscale (16): somatic concern, anxiety, guilt feelings, tension, mannerisms and posturing, depression, motor retardation, uncooperativeness, unusual thought content, disorientation, poor attention, lack of judgment and insight, disturbance of volition, poor impulse control, preoccupation, and active social avoidance). Severity was rated on 7-point scale with scores 1 (absence) & 7 (extremely severe). The PANSS Total score ranged from 7 (best possible outcome) to 210 (worst possible outcome).
Time Frame: From Baseline up to 52 Weeks including Week24, Week52, and Last Visit(LOCF)
Population: Efficacy sample（FAS : Full Analysis Set） consisted of all participants who received at least one dose of study medication and have Baseline and at least one Post-Baseline PANSS total score evaluation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | New Subjects | Rollover Subjects
Number analyzed (Participants) | 182 | 97
units on a scale
  Week24 | -5.31 (9.00) | -7.20 (12.59)
  Week52 | -7.01 (10.56) | -9.44 (15.16)
  Last Visit | -3.11 (12.76) | -2.58 (15.56)

3. Secondary Outcome: Mean Change From Baseline in PANSS Positive Subscale Score
Description: The PANSS consisted of three subscales that contained a total of 30 symptom constructs. For each symptom construct, severity is rated on a 7-point scale, with a score of 1 indicated the absence of symptoms and a score of 7 indicated extremely severe symptoms. In PANSS positive subscale, the 7 positive symptom constructs were: delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, and hostility. The PANSS positive subscale score ranged from 7 (best possible outcome) to 49 (worst possible outcome).
Time Frame: From Baseline up to 52 Weeks including Week24, Week52, and Last Visit(LOCF)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | New Subjects | Rollover Subjects
Number analyzed (Participants) | 182 | 97
units on a scale
  WEEK24 | -1.09 (2.27) | -1.53 (3.40)
  WEEK52 | -1.13 (2.73) | -1.61 (4.41)
  Last Visit | -0.19 (3.96) | 0.24 (4.83)

4. Secondary Outcome: Mean Change From Baseline in PANSS Negative Subscale Score
Description: The PANSS consisted of three subscales that contained a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 indicated the absence of symptoms and a score of 7 indicated extremely severe symptoms. In PANSS negative subscale the severity was rated for the following 7 negative symptom constructs: blunted affect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, stereotyped thinking. The PANSS negative subscale score ranged from 7 (best possible outcome) to 49 (worst possible outcome).
Time Frame: From Baseline up to 52 Weeks including Week24, Week52, and Last Visit(LOCF)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | New Subjects | Rollover Subjects
Number analyzed (Participants) | 182 | 97
units on a scale
  Week24 | -1.64 (3.22) | -1.49 (3.84)
  Week52 | -2.27 (3.85) | -2.02 (4.47)
  Last Visit | -1.43 (3.85) | -0.89 (3.92)

5. Secondary Outcome: Mean Change From Baseline in Clinical Global Impression-Severity of Illness (CGI-S)
Description: Severity of illness for each participant was rated using the CGI-S, which was the secondary efficacy endpoint. To perform this assessment, the study physician answered the following question: "Considering your total clinical experience with this particular population, how mentally ill is the participant at this time?" Response choices included: 0 = not assessed; 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants.
Time Frame: From Baseline up to 52 Weeks including Week24, Week52, and Last Visit(LOCF)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | New Subjects | Rollover Subjects
Number analyzed (Participants) | 182 | 97
units on a scale
  Week24 | -0.26 (0.71) | -0.20 (0.75)
  Week52 | -0.28 (0.67) | -0.15 (0.82)
  Last Visit | -0.13 (0.81) | 0.03 (0.92)

6. Secondary Outcome: Mean Clinical Global Impression - Global Improvement(CGI-I)
Description: The efficacy of trial medication was rated for each participant using the CGI-I. The study physician would rate the participant's total improvement whether or not it is due entirely to drug treatment. All responses were compared to the participant's condition at Baseline prior to the first dose of study medication. Response choices included: 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse.
Time Frame: From Baseline up to 52 Weeks including Week24, Week52, and Last Visit(LOCF)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | New Subjects | Rollover Subjects
Number analyzed (Participants) | 182 | 97
units on a scale
  Week24 | 3.09 (0.94) | 3.16 (0.90)
  Week52 | 3.09 (0.91) | 3.22 (0.99)
  Last Visit | 3.48 (1.22) | 3.86 (1.27)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from signing of the informed consent form until follow-up for up to 30 days after the completion of the treatment period (52 weeks).
Description: Incidence of Non-Serious TEAE of at Least 5% in Any Group by System Organ Class and MedDRA Preferred Term
Arm/Group | New Subjects | Rollover Subjects
All-Cause Mortality (participants affected / at risk) | 0/183 | 0/98
Serious Adverse Events (participants affected / at risk) | 19/183 | 18/98
Other Adverse Events (participants affected / at risk) | 112/183 | 50/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | New Subjects (N=183) | Rollover Subjects (N=98)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Meningitis aseptic (Infections and infestations) | 0 | 1
Heat illness (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Akathisia (Nervous system disorders) | 1 | 1
Extrapyramidal disorder (Nervous system disorders) | 1 | 0
Schizophrenia (Psychiatric disorders) | 17 | 13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | New Subjects (N=183) | Rollover Subjects (N=98)
Diarrhoea (Gastrointestinal disorders) | 10 | 3
Nasopharyngitis (Infections and infestations) | 46 | 19
Weight increased (Investigations) | 9 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 4
Akathisia (Nervous system disorders) | 15 | 7
Headache (Nervous system disorders) | 19 | 3
Somnolence (Nervous system disorders) | 13 | 3
Tremor (Nervous system disorders) | 4 | 8
Schizophrenia (Psychiatric disorders) | 21 | 13
Insomnia (Psychiatric disorders) | 15 | 2
Eczema (Skin and subcutaneous tissue disorders) | 5 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No